CLINICAL TRIAL: NCT00161603
Title: Cornell Translational Behavioral Science Research Consortium: Angioplasty Qualitative Study
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Mary E. Charlson, MD, Weill Cornell Medical College
Other Study IDs: N01-HC-25196 (0698-267); N01HC25196 (NIH)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Angioplasty Patients
Keywords: Angioplasty; Behavior change; Physical activity; Risk reduction
MeSH Terms: conditions — Motor Activity; Risk Reduction Behavior

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Semi-structured, open-ended interviews

SUMMARY:
To explore and illuminate the cultural, social, and psychological factors that either facilitate or serve as barriers to behavioral change in angioplasty patients. Through a series of open-ended questions we will explore and build a better understanding of how culturally different patient groups perceive heart disease and the difficulties in changing health behavior. In addition, we hope to better understand and anticipate barriers and issues that participants face in successfully changing their behaviors.

DETAILED DESCRIPTION:
1. To explore and illuminate the cultural, social, and psychological factors that either facilitate or serve as barriers to behavioral change in angioplasty patients. Through a series of open-ended questions we will explore and build a better understanding of how culturally different patient groups perceive heart disease and the difficulties in changing health behavior. In addition, we hope to better understand and anticipate barriers and issues that participants face in successfully changing their behaviors.
2. To use the responses obtained in the qualitative interviews to inform how we should operationalize and tailor the positive affect induction and self-affirmation intervention methods in each of the populations under study. Specifically, this involves assessing what small gifts participants prefer to receive and what would be most effective in inducing positive affect.

ELIGIBILITY:
Inclusion Criteria:

* Post-angioplasty patients who had previously participated in an RCT designed to motivate multi-behavior change.

Exclusion Criteria:

* Patients who refuse to be interviewed, Patients who were not enrolled in the parent trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2003-04; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- The New York Presbyterian Hospital-Weill Medical Center, New York, New York, United States

REFERENCES:
- [Result] Janey C. Peterson, RN, MA, Paul A. Pirraglia, MD, Sung Lee, MD, Laura Robbins, DSW, John P. Allegrante, PhD and Mary E. Charlson, MD. Living with heart disease: A qualitative study. Annals of Behavioral Medicine; 29(Supp), p. 28. April 14, 2005, Boston, MA.